CLINICAL TRIAL: NCT02415452
Title: Retinal Artery Lesions to Predict Long-term Outcomes in Patients With Acute Coronary Syndrome After Drug-Eluting Stent Implantation
Brief Title: Researches of Retinal Artery Lesions and Acute Coronary Syndrome
Acronym: REACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Mentougou District Hospital (Unknown); Beijing Haidian Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Beijing Tiantan Hospital, Capital Medical University
Other Study IDs: REACS
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome
Keywords: relationship; retinal artery lesions; long-term outcomes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Coronary Syndrome (ACS) patients: Acute coronary syndrome (ACS) patients who underwent coronary angiography ,drug-eluting stent (DES) implantation, and eye fundus examination.
  Interventions: Procedure: drug-eluting stent implantation

INTERVENTIONS:
Procedure: drug-eluting stent implantation — The DES contains Firebird , sirolimus-eluting stents, paclitaxel-eluting stents , or zotarolimus-eluting stents . Unfractionated heparin was used during percutaneous coronary intervention .A loading dose of 300 mg clopidogrel was given to all patients prior to PCI, followed by a maintenance dose of 75 mg daily for 12 months before it was stopped.
  Other Names: DES

SUMMARY:
This study is to investigate the relationship between staging of retinal artery lesions and the prognosis of acute coronary syndrome (ACS) in a Chinese population. All the patients were divided into four groups according retinal artery lesions.The endpoints were main adverse cardiovascular and cerebrovascular events (MACCE), including all-cause death, myocardial infarction (MI), and stroke after 3 to 6 years of follow-up.

DETAILED DESCRIPTION:
The aim of this study was to determine whether retinal artery lesions can predict long-term adverse outcomes in acute coronary syndrome (ACS) patients after drug-eluting stent (DES) implant.

A total of 660 consecutive patients with ACS who underwent coronary angiography and percutaneous coronary intervention enrolled this study at the Beijing Mentougou District Hospital, Beijing Tiantan Hospital and Beijing Shijitan Hospital. All the subjects were divided into two groups based on the retinal artery lesions: Group 1, retinal artery lesions≤ Stage 2 (n=296) and group 2 (n=364), retinal artery lesions > Stage 2. Beside,the eye fundus examination was done in all patients to mesure the extent and severity of atherosclerotic vascular lesions in the retinal arteries . Patients were excluded from the study if they had severe nephropathy (GFR< 30 mL/min/1.73 m2), vascular obstruction, acute illnesses or any other condition that was thought to contraindicated coronary angiography.

Primary endpoint was all-cause mortality. The composite endpoint was defined as major adverse cardiac and cerebrovascular events (MACCE), namely recurrent serious angina pectoris, nonfatal MI, revascularization and stroke.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with ACS who performed coronary angiography (CAG) and percutaneous coronary intervention (PCI).

Exclusion Criteria:

* Patients were excluded from the study if they had heart failure, malignancies, renal insufficiency (creatinine > 133µmol/L), liver disease, stroke and severe lung disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. acs patients in beijing mentougou district hospital
  2. acs patients in beijing shijitan hospital
  3. acs patients in beijing tiantan hospital
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2006-07; Primary Completion 2013-05 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Main cardiac events | July 1, 2006 to December 31, 2015, up to 9 years
  recurrent serious angina pectoris, nonfatal MI, revascularization and stroke

REFERENCES:
- [Result] Sharrett AR, Hubbard LD, Cooper LS, Sorlie PD, Brothers RJ, Nieto FJ, Pinsky JL, Klein R. Retinal arteriolar diameters and elevated blood pressure: the Atherosclerosis Risk in Communities Study. Am J Epidemiol. 1999 Aug 1;150(3):263-70. doi: 10.1093/oxfordjournals.aje.a009997. PMID 10430230
- [Result] Tedeschi-Reiner E, Strozzi M, Skoric B, Reiner Z. Relation of atherosclerotic changes in retinal arteries to the extent of coronary artery disease. Am J Cardiol. 2005 Oct 15;96(8):1107-9. doi: 10.1016/j.amjcard.2005.05.070. Epub 2005 Aug 29. PMID 16214446
- [Result] Cheung N, Bluemke DA, Klein R, Sharrett AR, Islam FM, Cotch MF, Klein BE, Criqui MH, Wong TY. Retinal arteriolar narrowing and left ventricular remodeling: the multi-ethnic study of atherosclerosis. J Am Coll Cardiol. 2007 Jul 3;50(1):48-55. doi: 10.1016/j.jacc.2007.03.029. Epub 2007 Jun 18. PMID 17601545
- [Result] Klein R, Sharrett AR, Klein BE, Chambless LE, Cooper LS, Hubbard LD, Evans G. Are retinal arteriolar abnormalities related to atherosclerosis?: The Atherosclerosis Risk in Communities Study. Arterioscler Thromb Vasc Biol. 2000 Jun;20(6):1644-50. doi: 10.1161/01.atv.20.6.1644. PMID 10845884
- [Result] SCHEIE HG. Evaluation of ophthalmoscopic changes of hypertension and arteriolar sclerosis. AMA Arch Ophthalmol. 1953 Feb;49(2):117-38. doi: 10.1001/archopht.1953.00920020122001. No abstract available. PMID 13007237
- [Result] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Result] Klein R, Klein BE, Knudtson MD, Wong TY, Cotch MF, Liu K, Burke G, Saad MF, Jacobs DR Jr. Prevalence of age-related macular degeneration in 4 racial/ethnic groups in the multi-ethnic study of atherosclerosis. Ophthalmology. 2006 Mar;113(3):373-80. doi: 10.1016/j.ophtha.2005.12.013. PMID 16513455
- [Result] Wong TY, Klein R, Islam FM, Cotch MF, Folsom AR, Klein BE, Sharrett AR, Shea S. Diabetic retinopathy in a multi-ethnic cohort in the United States. Am J Ophthalmol. 2006 Mar;141(3):446-455. doi: 10.1016/j.ajo.2005.08.063. PMID 16490489
- [Result] Shah A, Gnoj J, Fisher VJ. Complications of selective coronary arteriography by the Judkins technique and their prevention. Am Heart J. 1975 Sep;90(3):353-9. doi: 10.1016/0002-8703(75)90325-7. PMID 1163427
- [Result] Wong TY, Klein R, Sharrett AR, Duncan BB, Couper DJ, Tielsch JM, Klein BE, Hubbard LD. Retinal arteriolar narrowing and risk of coronary heart disease in men and women. The Atherosclerosis Risk in Communities Study. JAMA. 2002 Mar 6;287(9):1153-9. doi: 10.1001/jama.287.9.1153. PMID 11879113
- [Result] Wang L, Wong TY, Sharrett AR, Klein R, Folsom AR, Jerosch-Herold M. Relationship between retinal arteriolar narrowing and myocardial perfusion: multi-ethnic study of atherosclerosis. Hypertension. 2008 Jan;51(1):119-26. doi: 10.1161/HYPERTENSIONAHA.107.098343. Epub 2007 Nov 12. PMID 17998474
- [Result] Wang DZ, Tang Q, Hua Q. Prediction of coronary artery disease using pulse wave velocity and retinal artery lesions. Tohoku J Exp Med. 2011 Sep;225(1):17-22. doi: 10.1620/tjem.225.17. PMID 21841352
- [Result] Wong TY, Klein R, Sharrett AR, Couper DJ, Klein BE, Liao DP, Hubbard LD, Mosley TH; ARIC Investigators. Atheroslerosis Risk in Communities Study. Cerebral white matter lesions, retinopathy, and incident clinical stroke. JAMA. 2002 Jul 3;288(1):67-74. doi: 10.1001/jama.288.1.67. PMID 12090864
- [Result] Wong TY, Rosamond W, Chang PP, Couper DJ, Sharrett AR, Hubbard LD, Folsom AR, Klein R. Retinopathy and risk of congestive heart failure. JAMA. 2005 Jan 5;293(1):63-9. doi: 10.1001/jama.293.1.63. PMID 15632337
- [Result] Smith W, Wang JJ, Wong TY, Rochtchina E, Klein R, Leeder SR, Mitchell P. Retinal arteriolar narrowing is associated with 5-year incident severe hypertension: the Blue Mountains Eye Study. Hypertension. 2004 Oct;44(4):442-7. doi: 10.1161/01.HYP.0000140772.40322.ec. Epub 2004 Aug 9. PMID 15302843
- [Result] Ikram MK, Witteman JC, Vingerling JR, Breteler MM, Hofman A, de Jong PT. Retinal vessel diameters and risk of hypertension: the Rotterdam Study. Hypertension. 2006 Feb;47(2):189-94. doi: 10.1161/01.HYP.0000199104.61945.33. Epub 2005 Dec 27. PMID 16380526
- [Result] Wang JJ, Taylor B, Wong TY, Chua B, Rochtchina E, Klein R, Mitchell P. Retinal vessel diameters and obesity: a population-based study in older persons. Obesity (Silver Spring). 2006 Feb;14(2):206-14. doi: 10.1038/oby.2006.27. PMID 16571845
- [Result] Sellke FW, Armstrong ML, Harrison DG. Endothelium-dependent vascular relaxation is abnormal in the coronary microcirculation of atherosclerotic primates. Circulation. 1990 May;81(5):1586-93. doi: 10.1161/01.cir.81.5.1586. PMID 2110036
- [Result] Wu Y, Li S, Zu X, Du J, Wang F. Changes of central retinal artery blood flow and endothelial function in patients with coronary artery disease. Curr Eye Res. 2007 Sep;32(9):813-7. doi: 10.1080/02713680701572664. PMID 17882714